CLINICAL TRIAL: NCT05995262
Title: Effect of a Pharmacist-led, Collaborative Practice on Clinical Outcomes in Persons with Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 115.PHA.2022.C
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Diabetes; Type2diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HbA1c: Minimum of one HbA1c reading within 90 days prior to first visit AND one HgbA1c reading within 90 days after the last clinic encounter
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Data collection via retrospective chart review of patients from the Cedar Hill Clinic who had at least two visits with the clinical pharmacist between January 5, 2022 through December 31, 2022

SUMMARY:
Diabetes is a complex chronic illness known for its high prevalence (11.3% in the United States), significant healthcare burdens in terms of cost and management, and high mortality rate (seventh leading cause of death in the United States in 2019). Diabetes-related complications including ischemic heart disease, stroke, hyperglycemic crises, amputations, and hypoglycemia accounted for 8.25 million hospital discharges and 25.9% of emergency department visits, contributing towards the $327 billion total cost of diabetes in 2017. Proper treatment of diabetes is integral to reduce a patient's risk of developing complications; however, a number of barriers can create additional burdens for persons with diabetes.

Several studies have also demonstrated reductions in hospitalizations and/or ED visits for patients enrolled in pharmacist-led collaborative practice models. While the literature as a whole clearly describes the impact of ambulatory pharmacist intervention in achieving guideline-based clinical goals (i.e., HbA1c, blood pressure), few studies have reported on adherence with guideline-driven pharmacotherapy pre- and post-pharmacist intervention, or on pharmacist impact in reducing medication burden.

DETAILED DESCRIPTION:
Diabetes is a complex chronic illness known for its high prevalence (11.3% in the United States), significant healthcare burdens in terms of cost and management, and high mortality rate (seventh leading cause of death in the United States in 2019). Diabetes-related complications including ischemic heart disease, stroke, hyperglycemic crises, amputations, and hypoglycemia accounted for 8.25 million hospital discharges and 25.9% of emergency department (ED) visits, contributing towards the $327 billion total cost of diabetes in 2017. Proper treatment of diabetes is integral to reduce a patient's risk of developing complications; however, a number of barriers can create additional burdens for persons with diabetes (PWD). The root of these barriers affecting diabetes care is a topic of significant discussion especially given the emergence of conversations surrounding social determinants of health (SDOH) in recent years. A 2019 article from Annual Review of Public Health suggests that PWD experience health disparity, which are preventable differences in quality of healthcare and outcomes. This article discusses that health disparity is largely due to SDOH which are defined as the economic, environmental, political, and social conditions in which people live. Unfortunately, published research thus far has not identified strategies to reduce diabetes-related health inequity across the entire population. When providers recognize and discuss non-medical factors that influence PWD's health outcomes (e.g., food security, housing stability, transportation access, and financial security), they are able to promote health equity within their practice. Realistically, many providers have limited time to devote to individual patient encounters which often focus on immediate medical issues and eclipse discussions of non-medical issues, pharmacotherapy, and lifestyle changes. Thus, multidisciplinary care teams, including dieticians, nurses, and pharmacists, are recommended by the American Diabetes Association's (ADA) Standard of Care in Diabetes to ensure PWD receive the comprehensive care they need.

Within these teams, ambulatory care pharmacists are uniquely equipped to utilize their strong background in pharmacotherapy to provide chronic disease state medication management services for core primary care disease states, such as diabetes, hypertension, and hyperlipidemia. In many settings, ambulatory care pharmacists work under collaborative practice agreements (CPA), which are legal arrangements between pharmacists and physicians that allow for expanded services. The additional abilities granted within CPAs allow clinical pharmacists to assume professional responsibility by performing patient assessments, counseling, and referrals; ordering laboratory tests; administering drugs; and selecting, initiating, monitoring, continuing, and adjusting drug regimens. By allowing pharmacists to take on this prescribing role within a multidisciplinary team, patients receive more individualized, patient-centered care as recommended by ADA's Standard of Care in Diabetes and there is reduced clinical inertia (i.e., lack of treatment intensification in a patient not at evidence-based goals for care). In fact, patients receiving care from pharmacists under CPA were shown to have significantly better outcomes compared to patients receiving "usual care" without pharmacist intervention. Studies in a variety of ambulatory settings have illustrated that pharmacist intervention can significantly improve clinical outcomes in terms of hemoglobin A1C (HbA1c) level, blood pressure control, lipid panels, and body mass index. One study of a pharmacist-driven type 2 diabetes mellitus (T2DM)-targeted collaborative practice in an urban underserved clinic demonstrated significant improvements not only in HbA1c and tobacco cessation but also in guideline recommended utilization of statins and angiotensin-converting enzyme inhibitor/angiotensin receptor blockers. Several studies have also demonstrated reductions in hospitalizations and/or ED visits for patients enrolled in pharmacist-led collaborative practice models. While the literature as a whole clearly describes the impact of ambulatory pharmacist intervention in achieving guideline-based clinical goals (i.e., HbA1c, blood pressure), few studies have reported on adherence with guideline-driven pharmacotherapy pre- and post-pharmacist intervention, or on pharmacist impact in reducing medication burden.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Minimum of two visits with clinical pharmacist during 2022
* Minimum of one HbA1c reading within 90 days prior to first visit AND one HgbA1c reading within 90 days after the last clinic encounter

Exclusion Criteria:

* Clinic patients without diagnosis of type 1 diabetes mellitus or T2DM which, per ADA 2022 Standards of Care, is defined as an HbA1c of >6.5%

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minimum of one HbA1c reading within 90 days prior to first visit AND one HgbA1c reading within 90 days after the last clinic encounter
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c levels | within 90 days
  HbA1c will be evaluated within 90 days prior to the first visit and within 90 days after the last clinic encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Proffitt, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No